CLINICAL TRIAL: NCT03299907
Title: COPD MSA 3 Regions: Epidemiology and Risk Factors of COPD in Rural Environment (BPCO MSA 3Régions : épidémiologie et Facteurs de Risque de la BPCO en Milieu Rural)
Brief Title: COPD MSA 3 Regions: Epidemiology and Risk Factors of COPD in Rural Environment (BM3R)
Acronym: BM3R
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Mutualité sociale agricole (Unknown)
Responsible Party: Sponsor
Other Study IDs: P/2013/161
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Subject with FEV1/FVC post BD < 0.7 or LLN
  Interventions: Diagnostic Test: Spirometry
- Non COPD: Subject with FEV1/FVC post BD >= 0.7 or LLN
  Interventions: Diagnostic Test: Spirometry

INTERVENTIONS:
Diagnostic Test: Spirometry

SUMMARY:
The agricultural environment presents a unique profile in terms of epidemiology of pulmonary diseases. Certainly due to persistent exposure to organic particles, the prevalence of COPD is higher in farmers than in the general population, despite less smoking. It is likely that the risk of COPD depends on several factors, such as the type of farm, local conditions and the region where the farm is located. It is important to diagnose COPD at an early stage in order to initiate appropriate therapy, and implement secondary prevention with a view to limiting deterioration of respiratory function and reducing complications. In this context, the aims of BM3R project were: (1) to study the epidemiology of COPD in a large representative sample of French farmers, in order to identify the types of farming, working conditions and regions that are associated with the presence of COPD; and (2) to develop a score to identify patients at risk and optimise diagnosis of COPD in the context of a screening programme.

ELIGIBILITY:
Inclusion Criteria:

* > 40 years old and < 75 years old
* Affiliated to the MSA

Exclusion Criteria:

* COPD known

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data were collected between October 2012 and May 2013 in two French regions (Brittany and Franche-Comté) among affiliated members (farmers and administrative workers of both sexes) of the MSA.
Sampling Method: Non-Probability Sample
Enrollment: 5263 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2013-05-30 (Actual); Study Completion 2014-05-30 (Actual)

PRIMARY OUTCOMES:
FEV1/FVC | At the inclusion time

CONTACTS AND LOCATIONS:
Overall Officials: Bruno DEGANO, MD, Principal Investigator — CHU Besançon